CLINICAL TRIAL: NCT00129792
Title: Expectancy, Self-Efficacy and Outcomes in Metabolic Syndrome
Brief Title: Education, Counseling, and Drug Therapy to Reduce Symptoms of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U19AT002656 (NIH); U19AT002656-03 (NIH); U19AT002656-02 (NIH); U19AT002656 (NIH)
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Metabolic Syndrome X; Prediabetic State; Insulin Resistance; Obesity; Metabolic Diseases
Keywords: Blood Glucose; Cholesterol; Weight Loss; Insulin; Complementary Therapies
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State; Insulin Resistance; Obesity; Metabolic Diseases; Weight Loss | interventions — Dietary Supplements; Educational Status; Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Has 100% expectation of receiving supplement
  Interventions: Drug: Dietary supplement for weight loss; Behavioral: Education and counseling for weight loss
- 2 (Sham Comparator): Has 50% expectation of receiving supplement
  Interventions: Drug: Dietary supplement for weight loss; Behavioral: Education and counseling for weight loss
- 3 (Other): Has 0% expectation of receiving supplement.
  Interventions: Behavioral: Education and counseling for weight loss

INTERVENTIONS:
Drug: Dietary supplement for weight loss — The dietary supplement being investigated in this study is a natural product designed to reduce metabolic syndrome by decreasing hunger, increasing energy, and improving insulin function.
  Arms: 1; 2
Behavioral: Education and counseling for weight loss — Hour and a half weight loss education session weekly for 12 weeks.

SUMMARY:
This study will determine the effects of a supplement in reducing symptoms of metabolic syndrome, a collection of symptoms that increase the risk for developing heart disease, stroke, and diabetes.

DETAILED DESCRIPTION:
Metabolic syndrome is a serious condition involving abnormal glucose and lipid metabolism and obesity; these symptoms are associated with a two- to fourfold increased risk for cardiovascular disease and diabetes. The dietary supplement being investigated in this study is a natural product designed to reduce metabolic syndrome by decreasing hunger, increasing energy, and improving insulin function.

This study will last 12 weeks. Participants will be randomly assigned to one of three arms. Participants in Arm 1 will receive the supplement; participants in Arm 2 will have a 50% chance of receiving either the supplement or placebo; participants in Arm 3 will receive placebo. Participants will take their assigned pills 3 times daily for 12 weeks. A follow-up visit will occur at the end of the 12 weeks; there will be a debriefing visit shortly after the follow-up visit. Participants in all 3 arms will receive weekly education and counseling sessions on healthy lifestyle changes to encourage weight loss. Blood collection will occur at study start and at the end of 12 weeks for assessment of fasting blood glucose, insulin, cholesterol, and levels of certain hormones. Participants will also be asked to complete questionnaires at study entry and at Week 12; the questionnaires will assess depression, stress, self-absorption, optimism, food cravings, hunger, the degree to which participants seek pleasure from activities, and participants' thoughts about their ability to make behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 30 and 45
* Live in the Portland, Oregon metropolitan area
* Willing and able to complete a 12-week weight loss program
* Meet at least 3 of the following 5 criteria: 1) waist circumference greater than 40 inches for men and 35 inches for women; 2) fasting triglycerides higher than 150 mg/dl; 3) high density lipoprotein (HDL) lower than 40 mg/dl for men and 50 mg/dl for women; 4) systolic blood pressure (BP) of 130 mmHg or higher or diastolic BP of 85 mmHg or higher; 5) fasting glucose of 100 mg/dl or higher

Exclusion Criteria:

* Any medications, including dietary supplements, that could interfere with the study
* Medical conditions contraindicating a diet and exercise weight loss program
* History of congestive heart failure, stroke, myocardial infarction, coronary artery bypass graft, or atherosclerotic cardiovascular disease
* Current diagnosis of cancer
* Hospitalization for a psychiatric condition within 12 months prior to study entry
* Weight loss medications within 6 months prior to study entry
* Change in body weight greater than 5% within 6 months prior to study entry
* Consumption of more than 21 alcoholic drinks per week
* Current participation in another clinical trial OR living in the same household with another participant in this study
* Currently exercising for more than 30 minutes, 3 times per week
* Fasting blood glucose higher than 125 mg/dl
* BP higher than 145/90
* Triglycerides higher than 500 mg/dl
* Training as a health care provider or health scientist
* Pregnancy or breastfeeding

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cholesterol | baseline (Week 1) and outcome (Week 12)
insulin function | baseline (Week 1) and outcome (Week 12)
weight loss | baseline (Week 1) and outcome (Week 12)

SECONDARY OUTCOMES:
Cortisol levels | baseline (Week 1) and outcome (Week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Oken, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University General Clinical Research Center, Portland, Oregon, United States